CLINICAL TRIAL: NCT01932112
Title: Adenosine Effect on Persistent Pulmonary Vein Isolation Line Evaluation (APPLE Trial)
Acronym: APPLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, MD, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APPLE
Record Dates: First submitted 2013-08-14; First posted 2013-08-30 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Persistent Common Pulmonary Vein
Keywords: Pulmonary Vein Isolation; Adenosin effect; Atrial fibrillation ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adenosine arm (Other): single arm study
  Interventions: Drug: Adenosine arm

INTERVENTIONS:
Drug: Adenosine arm — After pulmonary vein isolation,20mg Intracardiac adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
  Other Names: APPLE

SUMMARY:
The investigators studied the effects of adenosine on the reconnection rate after successful pulmonary veins isolation by radiofrequency catheter ablation in patients with drug-resistant atrial fibrillation

DETAILED DESCRIPTION:
Pulmonary vein isolation has emerged as an effective therapy for paroxysmal atrial fibrillation. However, atrial fibrillation recurs in up to 50% of patients, generally because of recovery of pulmonary vein conduction.

Adenosine given during the initial procedure may reveal dormant pulmonary vein conduction, thereby identifying the need for additional ablation, leading to improved outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed atrial fibrillation
* recurrence of symptomatic atrial fibrillation in spite of Antiarrhythmic drug use
* written informed consent

Exclusion Criteria:

* intracardiac thrombus
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong seog Oh, MD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul st Mary's Hospital, Seoul, Seocho-Ku, South Korea

REFERENCES:
- [Derived] Kim JY, Kim SH, Song IG, Kim YR, Kim TS, Kim JH, Jang SW, Lee MY, Rho TH, Oh YS. Achievement of successful pulmonary vein isolation: methods of adenosine testing and incremental benefit of exit block. J Interv Card Electrophysiol. 2016 Sep;46(3):315-24. doi: 10.1007/s10840-016-0122-9. Epub 2016 Mar 9. PMID 26960977

RESULTS

PARTICIPANT FLOW:
Groups:
- Adenosine Arm: After pulmonary vein isolation, 20mg Iv adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
  Adenosine arm: After pulmonary vein isolation, 20mg Iv adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
Period: Overall Study
Arm/Group | Adenosine Arm
Started | 378
Completed | 378
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Adenosine Arm: After pulmonary vein isolation, 20mg Intracardiac adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
  Adenosine arm: After pulmonary vein isolation, 20mg Intracardiac adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
Arm/Group | Adenosine Arm
Number analyzed (Participants) | 378
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 255
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 378

OUTCOME MEASURES:

1. Primary Outcome: Reconnection of Pulmonary Vein Electrogram After Adenosine Infusion
Description: After pulmonary vein isolation, 20mg Intracardiac adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
Time Frame: 5 minutes after IV adenosine
Measure: Number; unit: participants
Groups:
- Adenosine Arm: After pulmonary vein isolation, 20mg Intracardiac adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
  Adenosine arm: After pulmonary vein isolation, 12mg Iv adenosine will be given to treatment group, will evaluate pulmonary vein reconnection.
Arm/Group | Adenosine Arm
Number analyzed (Participants) | 378
participants | 92

2. Secondary Outcome: Atrial Fibrillation Recurrence
Description: At 1 month, 3 month, 6 month and 12 months post ablation routine clinic visits, will perform electrocardiographically documented by electrogram (At 1,3,6,12 months post ablation) and Holter monitoring (At 12 months post ablation)
Time Frame: between 0 and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Adenosine Arm
Serious Adverse Events (participants affected / at risk) | 2/378
Other Adverse Events (participants affected / at risk) | 0/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adenosine Arm (N=378)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No